CLINICAL TRIAL: NCT04554602
Title: Fusion Ultrasound for Diagnosis and Monitoring of Endometriosis Lesions ENDOFUSION
Brief Title: Fusion Ultrasound for Diagnosis and Monitoring of Endometriosis Lesions
Acronym: ENDOFUSION
Status: Active, not recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP191069; 2019-A02828-49 (Other: IDRCB)
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient with endometriosis or suspicion of endometriosis: * Information and collection of the non-objection before inclusion
  * Interrogation, clinical examination, EHP30 and SF36 form at inclusion
  * MRI, pelvic ultrasound (coupled with fusion ultrasound)
  * Laparoscopy if indicated after MRI, ultrasound and fusion ultrasound
  * Monitoring by form and fusion ultrasound at 6 months and then once a year for 3 years
  Interventions: Diagnostic Test: Fusion ultrasound
- Patient with other gynaecological pathology: * Information and collection of the non-opposition before inclusion
  * Interrogation, clinical examination, EHP30 and SF36 form at inclusion
  * MRI, pelvic ultrasound (coupled with fusion ultrasound)
  * laparoscopy if indicated after MRI, ultrasound and fusion ultrasound
  Interventions: Diagnostic Test: Fusion ultrasound

INTERVENTIONS:
Diagnostic Test: Fusion ultrasound — Fusion ultrasound is a technique that allows a volume acquired in MRI to be coupled to an ultrasound scan with real-time image synchronisation.

SUMMARY:
The aim of the study is evaluate the fusion ultrasound performance compared to MRI and coelioscopy diagnosis when a surgical intervention is performed.

DETAILED DESCRIPTION:
The research is about diagnosis performance between fusion ultrasound and the gold standard (MRI coelioscopy ). Fusion ultrasound is a no-invasive scientific technical which allow with security to evaluate the progress of endometriosis lesions. During 39 months, 200 patients will be follow. In one arm, there is the control group with women without endometriosis. In the second arm, there is the patient with endometriosis. We will compare monitoring differences between gold standard and fusion ultrasound ( Cost assessment,exams duration, reproductibility, the link between symptoms and evolution of the lesion size).

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 50 years old
* Patient informed and who gave her non-opposition to participate in the research
* Patient with an indication for pelvic MRI and pelvic ultrasound either for the exploration of endometriosis or pelvic pain, or for another gynaecological pathology (ovarian cyst, poly-myomatous uterus, uterine malformation) outside of a proven cancer indication.
* Patient affiliated to a social security or entitled to a social security allowance

Exclusion Criteria:

* Patient with a proven cancerous pathology at the time of the prescription of the complementary examinations.
* Virgin patient
* Pregnant patient
* Patients under protective measures
* Contraindication to MRI (claustrophobia, intracorporeal metallic foreign body)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Any major patient with an indication for pelvic MRI and pelvic ultrasound outside a proven cancer indication (suspicion of endometriosis or other pathology for the control population).
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, positive predictive value (VPP) and negative predictive value (VPN) of fusion ultrasound compared to transvaginal ultrasound and MRI for the diagnosis of endometriosis lesions | 3 years and 3 months
  To evaluate the diagnostic performance of fusion ultrasound compared to transvaginal gynaecological ultrasound and MRI for the diagnosis of endometriosis lesions.

SECONDARY OUTCOMES:
Evaluate the reproducibility of the conclusions of the fusion ultrasound between 2 operators. | 3 years and 3 months
  Evaluation of the reproducibility by an intra-class correlation test for the conclusions of fusion ultrasound between two operators.
To evaluate the contribution of fusion ultrasound in the follow-up of patients suffering from endometriosis, in particular with an ultrasound follow-up in comparison with an initial reference MRI in the case of medical or surgical management. | 3 years and 3 months
  Correlation between the evolution of clinical and quality of life symptoms (EHP30 form and Short Form 36) and the evolution of lesion size between initial MRI and follow-up ultrasounds at 6 months and one year
Compare the duration of a standard ultrasound scan to an ultrasound scan with fusion | 3 years and 3 months
  Comparison of the average examination time by a Student T-test between standard and fusion ultrasound.
Evaluation of the cost of imaging for 3 years between an annual fusion ultrasound surveillance in replacement of a annual MRI surveillance | 3 years and 3 months
  Comparison of imaging costs will be carried out over 3 years between a conventional procedure with annual MRI and the procedure being evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Perrine CAPMAS, DR, Principal Investigator — APHP
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No